CLINICAL TRIAL: NCT06562192
Title: Phase I Open-label, Multi-center Study to Evaluate the Safety, Tolerability, Dosimetry, and Preliminary Activity of [177Lu]Lu-NNS309 in Patients With Pancreatic, Lung, Breast and Colorectal Cancers
Brief Title: Phase I Study of [177Lu]Lu-NNS309 in Patients With Pancreatic, Lung, Breast and Colorectal Cancers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CFXX489A12101; 2023-510356-23 (Other: CTIS)
Record Dates: First submitted 2024-08-16; First posted 2024-08-20 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Pancreatic Ductal Adenocarcinoma; Non-small Cell Lung Cancer; HR+/HER2- Ductal and Lobular Breast Cancer; Triple Negative Breast Cancer; Colorectal Cancer
Keywords: pancreatic ductal adenocarcinoma; non-small cell lung cancer; breast cancer; colorectal cancer; radioligand therapy (RLT); [177Lu]Lu-NNS309; [68Ga]Ga-NNS309
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Triple Negative Breast Neoplasms; Colorectal Neoplasms; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): Patients will receive [68Ga]Ga-NNS309, and if eligible, [177Lu]Lu-NNS309
  Interventions: Drug: [68Ga]Ga-NNS309; Drug: [177Lu]Lu-NNS309

INTERVENTIONS:
Drug: [68Ga]Ga-NNS309 — Radioligand imaging agent
Drug: [177Lu]Lu-NNS309 — Radioligand therapy

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, dosimetry and preliminary efficacy of [177Lu]Lu-NNS309 and the safety and imaging properties of [68Ga]Ga-NNS309 in patients aged ≥ 18 years with locally advanced or metastatic pancreatic ductal adenocarcinoma (PDAC), non-small cell lung cancer (NSCLC), HR+/HER2- ductal and lobular breast cancer (BC), triple negative breast cancer (TNBC) and colorectal cancer (CRC).

DETAILED DESCRIPTION:
The study will be done in two parts. The first part is called "escalation" and the second part is called "expansion". In both parts of the study, patients will initially be imaged with a [68Ga]Ga-NNS309 positron emission tomography (PET)/ computed tomography (CT) or PET/magnetic resonance imaging (MRI) scan and will be evaluated for eligibility for [177Lu]Lu-NNS309 treatment. In the escalation part, different doses of [177Lu]Lu-NNS309 will then be tested to identify recommended dose(s) (RD(s)) for further evaluation. The expansion part of the study will examine the safety and preliminary efficacy of [177Lu]Lu-NNS309 at the RD(s) determined during the escalation part. The end of study will occur when all patients per disease group in the expansion part have completed the follow-up for disease progression or discontinued from the study for any reason, and all patients have completed treatment and the 36-month long-term follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Patients with one of the following indications:
* Locally advanced unresectable or metastatic PDAC with disease progression following, or intolerance to cytotoxic chemotherapy, unless patient was ineligible to receive such therapy
* Locally advanced unresectable or metastatic NSCLC without any actionable genomic alterations with disease progression following, or intolerance to chemotherapy and immunotherapy, unless patient was ineligible to receive such therapy, or locally advanced unresectable or metastatic NSCLC with an actionable genomic alteration with disease progression following, or intolerance to targeted therapy, unless patient was ineligible to receive such therapy
* Locally advanced unresectable or metastatic HR+/HER2- ductal or lobular BC with disease progression following, or intolerance to, at least 2 lines of therapy, unless patient was ineligible to receive such therapy
* Locally advanced unresectable or metastatic TNBC with disease progression following, or intolerance to, at least 2 lines of therapy, unless patient was ineligible to receive such therapy
* (Dose escalation part only) Locally advanced or metastatic unresectable CRC with disease progression following, or intolerance to cytotoxic chemotherapy, unless patient was ineligible to receive such therapy. Patients with known microsatellite instability-high (MSI-H) or mismatch repair deficient (dMMR) status must also have had disease progression following, or intolerance to immune checkpoint inhibitor therapy, unless patient was ineligible to receive such therapy
* Patients must have lesions showing 68Ga-NNS309 uptake

Exclusion Criteria:

* Absolute neutrophil count (ANC) < 1.5 x 109/L, hemoglobin < 9 g/dL, or platelet count < 100 x 109/L
* QT interval corrected by Fridericia's formula (QTcF) ≥ 470 msec
* Creatinine clearance < 60 mL/min
* Unmanageable urinary tract obstruction or urinary incontinence
* Radiation therapy within 4 weeks prior to the first dose of [177Lu]Lu-NNS309

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2031-01-15 (Estimated); Study Completion 2031-01-16 (Estimated)

PRIMARY OUTCOMES:
Number of patients with dose limiting toxicities of [177Lu]Lu-NNS309 | From start of study treatment until 6 weeks or 4 weeks after, depending on dosing schedule
  A dose limiting toxicity (DLT) is defined as any adverse event or abnormal laboratory value of CTCAE (version 5.0) Grade 3 or higher that occurs within the DLT evaluation period and that is not primarily related to disease, disease progression, intercurrent illness, or concomitant medications with a few exceptions defined in the study protocol. Other clinically significant toxicities may be considered to be DLTs, even if not Grade 3 or higher.
Incidence and severity of adverse events and serious adverse events of [177Lu]Lu-NNS309 | From start of study treatment until completion of the 36 month follow up, assessed up to approximately 42 months
  The distribution of adverse events will be done via the analysis of frequencies for treatment-emergent adverse events (TEAEs) and serious adverse events (TESAEs) and through the monitoring of relevant clinical and laboratory safety parameters.
Dose modifications for [177Lu]Lu-NNS309 | From start of study treatment until last dose of study treatment, assessed up to approximately 24 weeks
  Dose modifications (dose interruptions and reductions) for [177Lu]Lu-NNS309 will be assessed and summarized using descriptive statistics. The number of patients with dose modification will be summarized by treatment groups.
Dose intensity for [177Lu]Lu-NNS309 | From start of study treatment until last dose of study treatment, assessed up to approximately 24 weeks
  Dose intensity for [177Lu]Lu-NNS309 will be assessed and summarized using descriptive statistics. Dose intensity is computed as the ratio of actual cumulative dose received and actual duration of exposure.

SECONDARY OUTCOMES:
Overall response rate (ORR) | Up to approximately 42 months
  ORR is defined as the proportion of patients with a BOR of complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 guidelines.
Duration of Response (DOR) | Up to approximately 42 months
  DOR is the time between the first documented response (CR or PR) and the date of progression according to RECIST v1.1 guidelines, or death due to any cause.
Disease control rate (DCR) | Up to approximately 42 months
  DCR is defined as the proportion of patients with a BOR of CR, PR or stable disease according to RECIST v1.1 guidelines.
Progression free survival (PFS) | Up to approximately 42 months
  PFS is defined as the time from the date of start of treatment to the date of the first documented progression according to RECIST v1.1 guidelines or death due to any cause.
Area Under the Curve (AUC) of [177Lu]Lu-NNS309 | Cycle 1 Day 1 (Pre-infusion, end of infusion, Post dose (30 minutes (min), 1 hours (hr), 2hr, 4hr, 6hr, 12hr)), Cycle 1 Day 2 (24hr), Cycle 1 Day 3 (48hr), Cycle 1 Day 4 (72hr), Cycle 1 Day 8 (168hr). The duration of a cycle is 4 weeks or 6 weeks.
  The [177Lu]Lu-NNS309 pharmacokinetic analysis will be performed based on decay-corrected blood radioactivity concentration data converted to mass units. AUC will be determined by non-compartmental methods.
Total body clearance of [177Lu]Lu-NNS309 | Cycle 1 Day 1 (Pre-infusion, end of infusion, Post dose (30 minutes (min), 1 hours (hr), 2hr, 4hr, 6hr, 12hr)), Cycle 1 Day 2 (24hr), Cycle 1 Day 3 (48hr), Cycle 1 Day 4 (72hr), Cycle 1 Day 8 (168hr). The duration of a cycle is 4 weeks or 6 weeks.
  The [177Lu]Lu-NNS309 pharmacokinetic analysis will be performed based on decay-corrected blood radioactivity concentration data converted to mass units. Total body clearance will be determined by non-compartmental methods.
Observed maximum blood concentration (Cmax) of [177Lu]Lu-NNS309 | Cycle 1 Day 1 (Pre-infusion, end of infusion, Post dose (30 minutes (min), 1 hours (hr), 2hr, 4hr, 6hr, 12hr)), Cycle 1 Day 2 (24hr), Cycle 1 Day 3 (48hr), Cycle 1 Day 4 (72hr), Cycle 1 Day 8 (168hr). The duration of a cycle is 4 weeks or 6 weeks.
  The [177Lu]Lu-NNS309 pharmacokinetic analysis will be performed based on decay-corrected blood radioactivity concentration data converted to mass units. Cmax will be determined by non-compartmental methods.
Observed maximum radioactivity concentration (Rmax) of [177Lu]Lu-NNS309 | Cycle 1 Day 1 (Pre-infusion, end of infusion, Post dose (30 minutes (min), 1 hours (hr), 2hr, 4hr, 6hr, 12hr)), Cycle 1 Day 2 (24hr), Cycle 1 Day 3 (48hr), Cycle 1 Day 4 (72hr), Cycle 1 Day 8 (168hr). The duration of a cycle is 4 weeks or 6 weeks.
  The [177Lu]Lu-NNS309 pharmacokinetic analysis will be performed based on decay-corrected blood radioactivity concentration data converted to mass units. Rmax will be determined by non-compartmental methods.
Volume of distribution (Vz) of [177Lu]Lu-NNS309 during the terminal phase | Cycle 1 Day 1 (Pre-infusion, end of infusion, Post dose (30 minutes (min), 1 hours (hr), 2hr, 4hr, 6hr, 12hr)), Cycle 1 Day 2 (24hr), Cycle 1 Day 3 (48hr), Cycle 1 Day 4 (72hr), Cycle 1 Day 8 (168hr). The duration of a cycle is 4 weeks or 6 weeks.
  The [177Lu]Lu-NNS309 pharmacokinetic analysis will be performed based on decay-corrected blood radioactivity concentration data converted to mass units. Vz will be determined by non-compartmental methods.
Terminal elimination half-life (T1/2) of [177Lu]Lu-NNS309 | Cycle 1 Day 1 (Pre-infusion, end of infusion, Post dose (30 minutes (min), 1 hours (hr), 2hr, 4hr, 6hr, 12hr)), Cycle 1 Day 2 (24hr), Cycle 1 Day 3 (48hr), Cycle 1 Day 4 (72hr), Cycle 1 Day 8 (168hr). The duration of a cycle is 4 weeks or 6 weeks.
  The [177Lu]Lu-NNS309 pharmacokinetic analysis will be performed based on decay-corrected blood radioactivity concentration data converted to mass units. T1/2 will be determined by non-compartmental methods.
Urinary excretion of radioactivity expressed as a percentage of injected dose (%ID) | Cycle 1: Pre-infusion, beginning of infusion to first SPECT/CT image acquisition, first SPECT/CT image acquisition to 6 hr post end of infusion (EOI), 6-24hr post EOI, 24-48hr post EOI, 48-72hr post EOI. The duration of a cycle is 4 weeks or 6 weeks.
  Urine elimination data for [177Lu]Lu-NNS309 will be assessed based on decay-corrected urine radioactivity concentration data. Urine elimination data will be expressed as percentage of injected dose (%ID).
Renal clearance of [177Lu]Lu-NNS309 | Cycle 1: Pre-infusion, beginning of infusion to first SPECT/CT image acquisition, first SPECT/CT image acquisition to 6 hr post end of infusion (EOI), 6-24hr post EOI, 24-48hr post EOI, 48-72hr post EOI. The duration of a cycle is 4 weeks or 6 weeks.
  Urine samples will be collected over specified time intervals and analyzed for radioactivity. Renal clearance of 177Lu-NNS309 will be summarized using descriptive statistics.
Absorbed dose of [177Lu]Lu-NNS309 | Cycle 1 Day 1, Cycle 1 Day 2 (24hr), Cycle 1 Day 3 (48hr), Cycle 1 Day 4 (72hr), Cycle 1 Day 8 (168hr). The duration of a cycle is 4 weeks or 6 weeks.
  Time activity curves (TACs) for the various organs and tumor lesions will be produced as fraction of injected activity per gram of tissue (%ID/g) as a function of time.
Incidence and severity of adverse events and serious adverse events of [68Ga]Ga-NNS309 | From Imaging visit until 3 days after 68Ga-NNS309 administration, assessed up to approximately 3 days.
  The distribution of adverse events will be done via the analysis of frequencies for TEAEs and TESAEs and through the monitoring of relevant clinical and laboratory safety parameters.
Visual and quantitative assessment of [68Ga]Ga-NNS309 uptake in normal tissues and tumor lesions over time | From 0 up to approximately 3 hrs after [68Ga]Ga-NNS309 dosing
  After [68Ga]Ga-NNS309 administration, [68Ga]Ga-NNS309 PET/CT or PET/MRI will be performed. Standardized uptake values (SUVs) of [68Ga]Ga-NNS309 in normal tissues and tumor lesions over time will be summarized.

CONTACTS AND LOCATIONS:
Locations (24):
- United States (8):
  - University of California LA, Los Angeles, California
  - Stanford University Medical Center, Palo Alto, California
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - BAMF Health, Grand Rapids, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Uni Of TX MD Anderson Cancer Cntr, Houston, Texas
  - University Of Washington, Seattle, Washington
- Novartis Investigative Site, Brussels, Belgium
- Canada (2):
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
- France (2):
  - Novartis Investigative Site, Bron
  - Novartis Investigative Site, Villejuif
- Germany (2):
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Rostock
- Novartis Investigative Site, Tel Aviv, Israel
- Italy (2):
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Reggio Emilia, RE
- Netherlands (2):
  - Novartis Investigative Site, Nijmegen, Gelderland
  - Novartis Investigative Site, Utrecht
- Spain (2):
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
- Switzerland (2):
  - Novartis Investigative Site, Geneva
  - Novartis Investigative Site, Lausanne

IPD SHARING:
Plan to Share IPD: No